CLINICAL TRIAL: NCT00517855
Title: A Phase 1 Double-Blind, Randomized, Placebo-Controlled, Single-Dose Escalation Study of the Safety and Pharmacokinetics of Intravenous Doses of PRTX-100 in Healthy Adult Subjects
Brief Title: Phase 1 Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of PRTX-100 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalex, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PRTX-100B-102
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Staphylococcal Protein A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: PRTX-100 (Staphylococcal protein A)

SUMMARY:
This study is the second human clinical study with PRTX-100. It is designed to assess the safety of a single intravenous (IV) dose of PRTX-100, as well as, how the drug is eliminated from the blood after dosing. Additionally, this study provides an opportunity to monitor immune system response to PRTX-100.

DETAILED DESCRIPTION:
A total of 20 healthy subjects will be enrolled into one of two dosing cohorts. Each dosing cohort will consist of 10 subjects. Within each cohort, subjects will be randomized to clinical trial material (CTM) (PRTX-100 or placebo) such that 8 subjects receive PRTX-100 and 2 subjects receive placebo. The PRTX-100 doses to be assessed in an ascending fashion are: 0.30 mcg/kg and 0.45 mcg/kg. Dosing of Cohort 2 will occur after the Investigator reviews Day 0-14 safety data and confers with the Sponsor Medical Monitor.

Subjects will be confined to the clinical pharmacology research unit for 5 days following dosing. Each cohort will have safety, pharmacokinetic, and pharmacodynamic assessments over the 5-day post-dose period. Subjects will also have follow-up assessments at 6, 7, 10 (±1), 14 (±1), 30 (±2), and 60 (±2) days post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written, informed consent
* Subjects in good health as determined by medical history, physical exam, standard safety laboratory tests, electrocardiogram (ECG) and vital signs
* Body Mass Index (BMI) within the range of 18.5-32 kg/m2
* Normotensive, defined as systolic blood pressure less than or equal to 150 mmHg and diastolic blood pressure less than or equal to 90 mmHg

Exclusion Criteria:

* Positive IgE anti-SpA titer on screening visit
* Male and female subjects unwilling to use acceptable forms of birth control throughout the study (acceptable forms include hormonal contraceptives used for at least 2 months prior to the screening visit, condom plus spermicide, cervical cap plus spermicide, diaphragm plus spermicide, or intrauterine device plus spermicide)
* Pregnant (β-hCG serum pregnancy test positive) or nursing (lactating) female subjects
* Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s), as determined by the investigator or designee
* Past medical history of deep venous thrombosis or thromboembolic disease, stroke, myocardial infarction, recurrent fetal loss, or prior diagnosis of Protein C deficiency or of factor V Leyden genotype
* Past history of vasculitis or autoimmune disease
* Clinical signs or symptoms of acute or resolving viral or bacterial infection
* History of atopic dermatitis or asthma
* History of current hepatitis or carriers of hepatitis B and/or hepatitis C (Hepatitis B surface antigen [HbsAg] positive or IgM antibodies to Hepatitis C [anti Hepatitis C IgM]).
* History of AIDS or determined HIV seropositive at screening
* Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs
* Clinically significant abnormalities in screening laboratory tests (hematology, chemistry, urinalysis)
* Positive urine drug test at screening or baseline (e.g., cocaine, amphetamines, barbiturates, opiates, benzodiazepines, etc.)
* Positive blood test for ethanol at screening or baseline
* Use of dietary supplements or prescription (with the exception of hormonal contraceptives), herbal, and over-the-counter medication(s) (with the exception of acetaminophen less than or equal to 1000 mg/day) within the 10 days prior to study Day 1
* Unable to refrain from tobacco or nicotine product use during the period of study confinement
* Donation of blood or plasma within 30 days prior to dosing
* Use of (an) investigational drug(s) within the 30 days or 5 half-lives (whichever is longer) prior to Day 1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Various timepoints over 14 days
Safety (assessed by adverse events, clinical lab tests, vital signs, ECG, physical exam) | Various timepoints over 60 days

SECONDARY OUTCOMES:
Immunogenicity | Various timepoints over 60days
Pharmacodynamic markers of drug effect | Various timepoints over 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Ballow, PharmD, Principal Investigator — Buffalo Clinical Research Center
Locations (1):
- Buffalo Clinical Research Center, Buffalo, New York, United States